CLINICAL TRIAL: NCT04850326
Title: A Randomized, Cross-Over Clinical Study to Evaluate the Acute Efficacy of AP Green Tea Extract After a Meal Composed of High-Fat/High-Carbohydrate
Brief Title: Clinical Study to Evaluate the Short Time Efficacy of AP Green Tea Extract Affer High Fat, High Carbohydrate Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amorepacific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: AP-R-2019-02
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Blood Glucose, High

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AP green tea extract (Experimental)
  Interventions: Dietary Supplement: AP green tea extract
- No intervention control (No Intervention)

INTERVENTIONS:
Dietary Supplement: AP green tea extract — single intake of AP green tea extract
  Arms: AP green tea extract

SUMMARY:
The objective of this clinical trial is to evaluate the short term effects of single dose AP green tea extracts in subjects with BMI (< 30 kg/m2) and fasting glucose level of > 100 mg/dL after high-fat/high-carbohydrate meal.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 19 years or over
* BMI < 30 kg/m2
* Fasting glucose level > 100 mg/dL (who is not under medication)
* Subjects who voluntarily decide to participate in this clinical study and sign the informed consent form on their own or through their representatives

Exclusion Criteria:

* At the screening visit, subjects who were diagnosed with obesity, diabetes, dyslipidemia and undergoing medication
* Subjects who were diagnosed with ventricular associated disease, unstable and uncontrolled chronic medical disease, hyper/hypothyroidism, or active malignant tumor and undergoing medication within 4 weeks prior to the first administration of the investigational product
* Subjects who have renal failure, acute or chronic hepatitis or known liver cirrhosis
* In addition to the above, subjects who are determined to be ineligible to participate in the clinical study according to the investigator's medical opinion

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2021-01-02 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
Change of Blood glucose level | 0 - 300 minute
  Change of Blood glucose level before and after high-carbohydrate/high-fat meal
Change of Insulin level | 0 - 300 minute
  Change of Insulin level before and after high-carbohydrate/high-fat meal
Change of Triglyceride level | 0 - 300 minute
  Change of Triglyceride level before and after high-carbohydrate/high-fat meal

CONTACTS AND LOCATIONS:
Locations (1):
- KangBuk Samsung Medical Center, Seoul, South Korea